CLINICAL TRIAL: NCT05464407
Title: Effekt af højproteindrik Med særligt Udvalgte næringsstoffer Til Mennesker Med Type 2 Diabetes og fodsår
Brief Title: High Protein Oral Nutritional Support With Special Nutrients in Patients With Type 2 Diabetes and Foot Ulcer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow patient reqruitment
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Randi Tobberup, Head of clinical dietitians, Ph.d., Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N20210057
Record Dates: First submitted 2022-04-22; First posted 2022-07-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Healing Ulcer

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cubitan (Experimental): 2 x oral nutritional supplement daily
  Interventions: Dietary Supplement: Cubitan
- Usual care (No Intervention): usual care

INTERVENTIONS:
Dietary Supplement: Cubitan — 2 bottles of Cubitan daily, for 12 weeks.
  Arms: Cubitan

SUMMARY:
To assess the supplement of a high protein oral nutritional supplement enriched with arginin, zink, vitamin c and antioxidants on the healing of foot ulcers in patients with type 2 diabetes mellitus

DETAILED DESCRIPTION:
The intervention group receive 2 x ONS drink daily (total 2 x 200 kcal, 3 g arginin, 250 ml vitamin C, 38 mg vitamin e, 64 micr.g selenium, 9 mg zink)

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes with newly diagnosed foot ulcer
* accept study participation

Exclusion Criteria:

* HbA1c >90 mmol/L
* cognitive challenges, fx dementia
* history with known alcohol or drug abuse
* allergy to milk or soya
* home less
* critical ischemia, distal blood pressure <0.30
* EGFR < 30
* dialysis or planned dialysis or patients with terminal kidney insufficiency

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
foot ulcer area | 12 weeks
  Reduction in ulcer area of the index ulcer, cm^2(based on height and width) within 12 weeks
Foot ulcer healing | 12 weeks
  Time to complete healing

SECONDARY OUTCOMES:
Compliance to intervention | 12 weeks
  number of bottles ingested/bottles expected to ingest
Accept of intervention | 12 weeks
  Measured by Visual Analogue Scale, minimum score 1, maximum score 5. Lower score is better outcome
HbA1c | 12 weeks and 6 months
  Change in HbA1c
Adverse events | 12 weeks and 6 months
  number of adverse events in relation to hypo- or hyperglycemia, amputations, kidney function
Body weight | 12 weeks and 6 months
  change in body weight
Improvement in Quality of life | 12 weeks and 6 months
  World Health Organisation - Five Well-Being Index (WHO 5). The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Number of foot ulcers | 12 weeks and 6 months
  number of foot ulcers
Depth foot ulcer | 12 weeks
  Reduction in depth within 12 weeks
Classifying/scoring of food ulcer | 12 weeks and 6 months
  Use of SINBAD (site-ischemia-neuropathy-bacterial infection-area-depth) score system. Minimum score 0, maximum score 6. Lower score is better outcome
Time to complete healing of foot ulcer | 6 months
  Time to complete healing of foot ulcer
  Time to complete heling of foot ulcer
Reduction in ulcer area | 6 months
  Reduction in ulcer area of the index ulcer, cm^2 (based on height and width)
Number of new foot ulcers | 12 weeks and 6 months
  Counting the number of new foot ulcers occuring after study inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Randi Tobberup, phd, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No